CLINICAL TRIAL: NCT07088653
Title: Clinical Evaluation of 0.12% Chlorhexidine Versus MicroRepair® ABX Mouthwash in the Non-Surgical Management of Plaque-Induced Gingivitis: A Randomized Controlled Trial
Brief Title: Comparison of 0.12% Chlorhexidine and MicroRepair ABX Mouthwash in Gingivitis Management
Acronym: GEM-CHX012
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-CHX0.12vsABX
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Gingivitis; Dental Plaque; Gingival Inflammation
Keywords: Chlorhexidine 0.12%; MicroRepair ABX; Gingivitis; Dental Plaque; Gingival Inflammation; Mouthwash; Oral Hygiene; Guided Biofilm Therapy; aMMP-8; Randomized Controlled Trial
MeSH Terms: conditions — Gingivitis; Dental Plaque | interventions — Chlorhexidine; Mouthwashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MicroRepair® ABX Mouthwash Group (Experimental): Participants will receive baseline clinical assessments (T0) and instructions for home oral hygiene. They will start a 14-day twice-daily regimen with MicroRepair® ABX mouthwash, containing zinc-hydroxyapatite and antibacterial agents. All participants will use a standardized sodium lauryl sulfate (SLS)-free toothpaste (Biorepair®). At the 1-month visit (T1), they will undergo professional supragingival prophylaxis with Guided Biofilm Therapy (GBT), including plaque disclosure, ultrasonic scaling (EMS Piezon), and air polishing with glycine powder. At 3 (T2) and 6 months (T3), GBT and the home mouthwash regimen will be repeated only if the Full Mouth Bleeding Score (FMBS) remains >10%.
  Interventions: Drug: MicroRepair ABX mouthwash
- 0.12% Chlorhexidine Mouthwash Group (Active Comparator): Participants will receive baseline clinical assessments (T0) and instructions for home oral hygiene. They will start a 14-day twice-daily regimen with 0.12% chlorhexidine (CHX) mouthwash. All participants will use the same standardized SLS-free toothpaste (Biorepair®). At the 1-month visit (T1), they will undergo professional supragingival prophylaxis with GBT, including plaque disclosure, ultrasonic scaling (EMS Piezon), and air polishing with glycine powder. At 3 (T2) and 6 months (T3), GBT and the home mouthwash regimen will be repeated only if FMBS remains >10%.
  Interventions: Drug: Chlorhexidine 0.12% mouthwash

INTERVENTIONS:
Drug: MicroRepair ABX mouthwash — Participants begin at T0 (baseline) with clinical assessments, oral hygiene instruction, and the start of a 14-day home regimen using MicroRepair® ABX mouthwash. The formulation contains zinc-hydroxyapatite with antibacterial agents (cetylpyridinium chloride, magnolol, honokiol). Mouthwash is used twice daily (10 mL for 30 seconds) without rinsing, and participants avoid food or drink for 1 hour afterward. All participants use the same sodium lauryl sulfate (SLS)-free toothpaste (Biorepair®) throughout the study.
  Other Names: MicroRepair® ABX
  Arms: MicroRepair® ABX Mouthwash Group
Drug: Chlorhexidine 0.12% mouthwash — Participants begin at T0 (baseline) with clinical assessments, oral hygiene instruction, and the start of a 14-day home regimen using 0.12% chlorhexidine (CHX) mouthwash. Mouthwash is used twice daily (10 mL for 30 seconds) without rinsing, and participants avoid food or drink for 1 hour afterward. All participants use the same SLS-free toothpaste (Biorepair®) throughout the study.
  Other Names: Chlorhexidine 0.12%
  Arms: 0.12% Chlorhexidine Mouthwash Group

SUMMARY:
This study is designed to compare two mouthwashes used after professional dental cleaning in patients with gingivitis, a common form of gum inflammation caused by dental plaque. The two mouthwashes being studied are 0.12% chlorhexidine (CHX), which has been widely used for many years, and MicroRepair® ABX, a newer biomimetic hydroxyapatite mouthwash.

All participants will receive the same professional cleaning using the Guided Biofilm Therapy (GBT) protocol. They will then be randomly assigned to use one of the two mouthwashes twice daily for 14 days. The study will measure improvements in gum health, including reduced inflammation and plaque, and will also look at possible side effects such as tooth staining and changes in taste. Other periodontal health measures and a salivary biomarker of inflammation (active matrix metalloproteinase-8, aMMP-8) will also be assessed.

Participants will be followed for 6 months. The results will help determine whether MicroRepair® ABX can provide an effective and well-tolerated alternative to chlorhexidine for managing gingivitis.

DETAILED DESCRIPTION:
Gingivitis is the most common reversible form of periodontal disease, caused primarily by bacterial biofilm accumulation along the gingival margin. Chlorhexidine digluconate has long been considered the gold standard adjunct to professional oral hygiene, but its prolonged use is associated with adverse effects such as tooth staining, taste alteration, and mucosal irritation. In recent years, biomimetic hydroxyapatite-based rinses (MicroRepair® ABX) have been proposed as a well-tolerated alternative with antibacterial, remineralizing, and potential anti-inflammatory properties.

This randomized, controlled, monocentric clinical trial aims to compare the clinical and biological effectiveness of a biomimetic hydroxyapatite mouthwash (MicroRepair® ABX) versus 0.12% chlorhexidine (CHX) in patients with generalized gingivitis. Forty adult patients will be randomly assigned to receive either professional oral hygiene followed by 14 days of adjunctive use of MicroRepair® ABX mouthwash, or professional oral hygiene followed by 14 days of 0.12% CHX rinse.

The primary endpoint is the reduction of probing pocket depth (PPD). Secondary outcomes include changes in gingival bleeding assessed by the Full Mouth Bleeding Score (FMBS), dental plaque accumulation assessed by the Full Mouth Plaque Score (FMPS), clinical attachment level (CAL), gingival recession (REC), salivary levels of active matrix metalloproteinase-8 (aMMP-8), tooth staining assessed by the Lobene Stain Index, dentinal hypersensitivity assessed by the Schiff Air Index, and patient-reported taste alterations.

Patients will be followed up at 2 weeks, 1 month, 3 months, and 6 months. This study is designed to generate novel evidence on whether biomimetic hydroxyapatite can provide a clinically effective and better-tolerated alternative to chlorhexidine in the management of gingivitis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 70 years
* Presence of generalized plaque-induced gingivitis (FMBS ≥ 25%, PPD ≤ 3 mm in ≥90% of sites)
* At least 20 natural teeth
* Good general health (ASA I or II)
* Signed written informed consent
* Willingness to comply with study protocol and attend all follow-up visits

Exclusion Criteria:

* Periodontitis (defined as interdental CAL ≥1 mm at ≥2 non-adjacent teeth)
* Systemic diseases affecting periodontal status (e.g., diabetes, immunodeficiencies)
* Antibiotic or anti-inflammatory therapy in the last 3 months
* Professional dental cleaning in the past 3 months
* Pregnancy or breastfeeding
* Known allergy to chlorhexidine or microRepair® components
* Use of orthodontic appliances or removable prostheses
* Smoking more than 10 cigarettes per day
* Participation in other clinical trials in the past 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Change in periodontal probing depth assessed by Probing Pocket Depth (PPD) | Baseline (T0), 2 weeks (T1), 1 month (T2), 3 months (T3), 6 months (T4)
  Periodontal probing depth (PPD) is defined as the distance from the gingival margin to the bottom of the gingival sulcus or periodontal pocket, measured in millimeters using a calibrated periodontal probe (Hu-Friedy PCP UNC 15). PPD is assessed at six sites per tooth (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, distolingual). For each participant, a mean PPD value is calculated at each time point. Typical scores range from 1 mm (healthy sulcus) to ≥7 mm (advanced pocket), with higher values indicating more severe periodontal inflammation or attachment loss.
  The primary endpoint is the change in mean PPD from baseline (T0) to 6 months (T4), comparing the two intervention groups: MicroRepair® ABX mouthwash regimen versus 0.12% chlorhexidine (CHX) mouthwash regimen.

SECONDARY OUTCOMES:
Change in plaque accumulation assessed by Full Mouth Plaque Score (FMPS) | Baseline (T0), 2 weeks (T1), 1 month (T2), 3 months (T3), 6 months (T4)
  The Full Mouth Plaque Score (FMPS) quantifies the percentage of tooth surfaces with visible dental plaque, assessed after plaque disclosure at four sites per tooth (mesial, buccal, distal, lingual). The score is calculated as the number of plaque-positive sites divided by the total number of sites ×100. Scores range from 0% (no plaque) to 100% (plaque on all surfaces). Lower scores indicate better oral hygiene. FMPS will be compared between groups across time points.
Change in gingival inflammation assessed by Full Mouth Bleeding Score (FMBS) | Baseline (T0), 2 weeks (T1), 1 month (T2), 3 months (T3), 6 months (T4)
  FMBS measures the percentage of bleeding sites after gentle probing at four sites per tooth (mesial, buccal, distal, lingual). It reflects the presence and severity of gingival inflammation. Scores range from 0% (no bleeding) to 100% (bleeding at all sites). A higher FMBS indicates more severe gingival inflammation. Comparison of FMBS over time will be used to assess clinical response to treatment.
Change in salivary inflammation assessed by activated Matrix Metalloproteinase-8 (aMMP-8) levels | Baseline (T0), 2 weeks (T1)
  Active matrix metalloproteinase-8 (aMMP-8) is a salivary biomarker of periodontal inflammation, measured with a commercial immunoenzymatic test (aMMP-8 Test®, Biomolecular Diagnostic). Results are expressed in nanograms per milliliter (ng/mL). Reference ranges: <8 ng/mL = no inflammation; 9-19 ng/mL = mild inflammation; ≥20 ng/mL = severe inflammation. aMMP-8 levels will be compared between groups from baseline (T0) to 2 weeks (T1).
Change in gingival recession assessed by Recession (REC) | Baseline (T0), 2 weeks (T1), 1 month (T2), 3 months (T3), 6 months (T4)
  Gingival Recession (REC) is defined as the distance in millimeters between the cemento-enamel junction (CEJ) and the gingival margin, measured at six sites per tooth with a calibrated periodontal probe. Scores typically range from 0 mm (no recession) to ≥5 mm (advanced recession). Higher values indicate greater apical migration of the gingival margin. REC will be compared between groups across time points.
Change in clinical attachment level assessed by Clinical Attachment Level (CAL) | Baseline (T0), 2 weeks (T1), 1 month (T2), 3 months (T3), 6 months (T4)
  Clinical Attachment Level (CAL) is the distance from the cemento-enamel junction (CEJ) to the bottom of the gingival sulcus or periodontal pocket, measured in millimeters at six sites per tooth with a calibrated periodontal probe (Hu-Friedy PCP UNC 15). Scores typically range from 0 mm (healthy attachment) to ≥7 mm (severe attachment loss). Higher values indicate more severe periodontal damage. CAL will be compared between groups across time points.
Change in extrinsic staining assessed by Lobene Stain Index Modified | Baseline (T0), 2 weeks (T1), 1 month (T2), 3 months (T3), 6 months (T4)
  The Modified Lobene Stain Index assesses extrinsic tooth staining on buccal and lingual/palatal surfaces. Each surface is scored for stain area and intensity, with total scores ranging from 0 (no stain) to 3 (severe stain). Higher scores indicate more pronounced extrinsic discoloration. Index scores will be compared between groups across time points.
Change in dentin hypersensitivity assessed by Schiff Air Index | Baseline (T0), 2 weeks (T1), 1 month (T2), 3 months (T3), 6 months (T4)
  The Schiff Air Index measures dentinal hypersensitivity in response to an air stimulus applied to the cervical area of the tooth. Scores range from 0 (no response) to 3 (painful response and request to stop). Higher scores indicate greater dentinal hypersensitivity. Scores will be compared between groups across time points.
Change in taste perception assessed by a validated taste alteration questionnaire | 2 weeks (T1), 1 month (T2), 3 months (T3), 6 months (T4)
  Taste perception will be evaluated using a validated patient-reported questionnaire that explores the presence and severity of taste alterations (e.g., bitter, metallic, or unpleasant taste). Each item is scored on a 5-point Likert scale: 0 = no alteration, 1 = mild alteration, 2 = moderate alteration, 3 = severe alteration, 4 = very severe alteration. The total score reflects the degree of dysgeusia perceived by the patient. Mean scores will be compared between groups at each time point to assess tolerability of the mouthwashes.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, Associate Professor, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the corresponding authors.